CLINICAL TRIAL: NCT02483598
Title: Mechanistic Investigation Of Intestinal Cytochrome p450 3A4 Following Roux-en-Y Surgery And Its Effect on Plasma Concentrations of Buspirone
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Initial analysis of results warranted a study re-design and work on the study was suspended.
Sponsor: North Dakota State University (Other)
Collaborators: Neuropsychiatric Research Institute, Fargo, North Dakota (Other)
Responsible Party: Principal Investigator, Kristine Steffen, Associate Professor, North Dakota State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: bus-000
Record Dates: First submitted 2015-06-22; First posted 2015-06-29 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Gastric Bypass
Keywords: buspirone; pharmacokinetics; Cytochrome P450 3A4
MeSH Terms: interventions — Buspirone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buspirone (Experimental): Buspirone alone
  Interventions: Drug: Buspirone; Drug: Buspirone and Grapefruit Juice
- Buspirone plus grapefruit juice (Active Comparator): Buspirone plus grapefruit juice
  Interventions: Drug: Buspirone; Drug: Buspirone and Grapefruit Juice

INTERVENTIONS:
Drug: Buspirone — The primary aim of this study is to compare the relative difference between the area-under-the-curve (AUC) of buspirone alone (buspirone) with the AUC of buspirone in the presence of grapefruit juice (buspirone + GFJ) in patients who underwent RYGB 9-18 months prior versus a control group of participants who have not undergone bariatric surgery.
Drug: Buspirone and Grapefruit Juice — Grapefruit juice will be given before and during buspirone administration to inhibit intestinal CYP3A4.

SUMMARY:
This study is to compare intestinal Cytochrome P450 3A4 (CYP3A4) activity in 9-18 month post weight loss surgery Roux-en-Y Gastric Bypass (RYGB) versus control subjects who have not had a weight loss surgery and are of similar age, gender, body mass index as the gastric bypass group. For this purpose, we will compare post-bariatric surgery patients with control subjects on alterations in systemic exposure of buspirone, a CYP3A4 substrate, when administered with grapefruit juice, a selective intestinal CYP3A4 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Age 18-65 (inclusive, at time of informed consent)
3. No tobacco use in the past three months.
4. Underwent Roux-en-Y Gastric Bypass weight loss surgery 9-18 months prior to study OR has not had a weight loss surgery but matches the gastric bypass patients on age, gender, and BMI.
5. Ability to read, write and understand English.
6. Expresses the ability/willingness to consume grapefruit juice.

Exclusion Criteria:

1. Taking a medication that has a clinically significant interaction with buspirone or grapefruit juice or an interaction that may alter the study data.
2. Hypersensitivity to buspirone or any excipient contained within the dosage forms or grapefruit juice.
3. Inability to tolerate repeated blood draws.
4. Any history of bipolar disorder or a psychotic disorder.
5. Current major depressive disorder or current suicidality.
6. Alcohol or substance dependence in the past year.
7. Currently pregnant or lactating or unwillingness to use medically accepted contraception during study.
8. Taking a medication which significantly alters gastrointesinal transit time.
9. Medical conditon which may increase participant risk with buspirone or grapefruit juice.
10. Self reported history of viral hepatits or HIV.
11. Positive urine drug screen unless documented prescription of a non-interacting medication.
12. Renal impairment as evidenced by an estimated glomerular filtration rate (eGFR) of less than or equal to 60 ml/min/1.73 m2 or other abnormality on a renal panel that the medical provider feels puts the participant at risk.
13. Hepatic insufficiency as defined by any hepatic enzyme greater than 3x the upper limit of normal or other hepatic laboratory abnormalities at the discretion of the medical provider.
14. Any contraindication to bioelectrical impedance analysis (BIA) such as pregnancy, the presence of a pacemaker or other implanted mechanical device.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Area-under-the-curve | 9-18 months following RYGB
  The primary aim of this study is to compare the relative difference between the area-under-the-curve (AUC) of buspirone alone (buspirone) with the AUC of buspirone in the presence of grapefruit juice (buspirone + GFJ) in patients who underwent RYGB 9-18 months prior versus a control group of participants who have not undergone bariatric surgery.

SECONDARY OUTCOMES:
Composite of pharmacokinetic measures compared between buspirone and buspirone with grapefruit juice in participants who have undergone RYGB and nonsurgical control participants. | 9-18 months following RYGB
  General pharmacokinetic comparisons (Cmax, Tmax, half-life, etc.) will be made between the two conditions.
Compare GLP-2 levels between the buspirone and buspirone with grapefruit juice in participants who have undergone RYGB and nonsurgical control participants. | 9-18 months following RYGB
  To compare GLP-2 levels between participants and drug conditions.